CLINICAL TRIAL: NCT00498771
Title: Aquatic Exercise Study for Breast Cancer Patients With Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 006-116
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Lymphedema
Keywords: Lymphedema; Aquatic Exercise; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aquatic Exercise arm (Active Comparator): Participants will attend 12 classes of aquatic exercise program (2-3 classes/weekly). Each one hour class is held in warm water pool which is 89 degrees and 3.5'-4'deep.Classes include low impact, dynamic movements for warm up, stretching and breathing exercises, upper and lower body resistance training, and cool down activities. Participants will be evaluated for Circumference & volumetric measurement of the affected limb, BMI, weight and height at the baseline, at 3rd week and at 6th week. Participant will complete a quality of life survey (QOL)at baseline, 6 week, 6 and 12 month.
  Interventions: Behavioral: Aquatic Exercise arm
- Control - No Exercise Arm (No Intervention): No exercise will be performed in Control arm. Participants will be evaluated for Circumference & volumetric measurement of the affected limb, BMI, weight and height at the baseline, at 3rd week and at 6th week. Participant will complete a quality of life survey (QOL) at baseline, 6 week, 6 and 12 month.

INTERVENTIONS:
Behavioral: Aquatic Exercise arm — Participants will attend 12 classes of aquatic exercise program (2-3 classes/weekly). Each one hour class is held in warm water pool which is 89 degrees and 3.5'-4'deep.Classes include low impact, dynamic movements for warm up, stretching and breathing exercises, upper and lower body resistance training, and cool down activities. Participants will be evaluated for Circumference & volumetric measurement of the affected limb, BMI, weight and height at the baseline, at 3rd week and at 6th week. Participant will complete a quality of life survey (QOL)at baseline, 6 week, 6 and 12 month.
  Arms: Aquatic Exercise arm

SUMMARY:
The purpose of this study is to determine what effects aquatic exercise has on participants with Lymphedema.

DETAILED DESCRIPTION:
This pilot study will examine the effectiveness of aquatic exercise in reducing Lymphedema. The study is designed for breast cancer patients who have developed Lymphedema following cancer treatment. Potential study participants should have explored conventional treatments such as decongestive therapy and lymph drainage massage before joining the study.

There are two groups that the participants may choose from until enrollment for the group has reached its capacity.The active arm of the study will attend 12 one-hour aquatic exercise classes and classes will be held in an indoor heated pool. There is no cost to the participants.Both the active arm and the control group (not attending aquatic exercise classes) will have 3 measurement assessments that will compare the circumference and volumetric measurement of arms, as well as height, weight and body mass index (BMI).

Both group will fill out a program questionnaire. Quality of life survey taken at baseline, week 6, month 6 and 12 will be compared. A follow up questionnaire will be completed at 6 and 12 month intervals, and annually for five years.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with Lymphedema
* Patients must have received standard Lymphedema treatment (Complete Decongestive Therapy) prior to participating in the study.
* Patients undergoing treatment will require written permission from their physician
* Complete an assessment by a licensed physical therapist before beginning the exercise program
* Patients must sign a consent form to participate

Exclusion Criteria:

* Patients undergoing treatment without physician's written permission
* Patients with health problems that contraindicate exercise
* Patients are not eligible if the physical therapy assessment identifies a contraindication to participation

Inclusion of Women and Minorities:

- Men, women and minorities with breast cancer related lymphedema are eligible

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-07; Primary Completion 2009-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Reduction of Lymphedema | baseline, week 6, month 6, and month 12
  Comparison of the circumference and volumetric measurements of the affected limb will be made prior to, midpoint and at completion of the 12 class program. Quality of life surveys taken at baseline, week 6, month 6 and 12 will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grant, M.D., Principal Investigator — Baylor Sammons Breast Center
Locations (1):
- Baylor Sammons Breast Center, Dallas, Texas, United States